CLINICAL TRIAL: NCT00569504
Title: Prevalence of the Metabolic Syndrome in Patients With Schizophrenia Taking Antipsychotics
Brief Title: Prevalence of the Metabolic Syndrome in SPR Taking Antipsychotics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National Hospital (Other Government)
Collaborators: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Shi Hyun Kang, Seoul National Hospital
Other Study IDs: snh001; PMSPSTA
Record Dates: First submitted 2007-12-06; First posted 2007-12-07 (Estimated); Last update posted 2009-06-12 (Estimated); Status verified 2009-06

CONDITIONS: Metabolic Syndrome; Schizophrenia
Keywords: schizophrenia; antipsychotics; metabolic syndrome; prevalence
MeSH Terms: conditions — Metabolic Syndrome; Schizophrenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood sampling
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A, observatoin: inpatients and outpatients in Seoul National Hospital

SUMMARY:
The purpose of this study is to assess the cross-sectional prevalence of the metabolic syndrome in patients with schizophrenia taking antipsychotics.

DETAILED DESCRIPTION:
Schizophrenic patients taking any kind of antipsychotics for at least 1 year at the Seoul National Hospital will be participated in this study.

we are planning to enroll approximately 1000 patients with schizophrenia.

For each subject

* abdominal circumference
* body mass index
* lipid profile : TG, HDL-chlo, total chol
* systolic/diastolic blood pressure
* fasting blood glucose will be measured.

we will calculate the rates of patients who meet the criteria for the Metabolic syndrome.

1. Abdominal obesity : absolute criteria
2. 2 or more of followings

   1. Triglyceride ≥ 150mg/dL or ongoing treatment
   2. HDL-cholesterol < 40mg/dL (men) HDL-cholesterol < 50mg/dL (female) or ongoing treatment
   3. Hypertension 130mmHg ≥ systolic 85mmHg ≥ diastolic or ongoing treatment
   4. FBS ≥ 100mg/dL or previous diagnosis of type II DM

ELIGIBILITY:
Inclusion Criteria:

* Patients taking a same antipsychotics at least more than one year
* schizophrenia or schizoaffective disorder

Exclusion Criteria:

* none

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: DSM-IV diagnosis of schizophrenia
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2007-12; Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
metabolic syndrome | cross-sectional

SECONDARY OUTCOMES:
each factor of metabolic syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Jong-il Lee, M.D., Study Director — Seoul National Hospital
Locations (1):
- Seoul National Hospital, Seoul, South Korea